CLINICAL TRIAL: NCT02584595
Title: An Evaluation of Inducible Monomorphic Ventricular Tachycardia (MMVT) in Patients With St. Jude Medical Implantable Cardioverter Defibrillator (ICD) Systems or Cardiac Resynchronization Therapy Defibrillation (CRT-D) Systems.
Brief Title: Evaluation of Inducible Monomorphic Ventricular Tachycardia (MMVT) in Patients With St. Jude Medical (SJM) Implantable Cardioverter Defibrillator (ICD) Systems or Cardiac Resynchronization Therapy Defibrillation (CRT-D) Systems.
Acronym: EPIC
Status: Withdrawn | Type: Observational
Why Stopped: Business decision
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10068
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Monomorphic Ventricular Tachycardia
Keywords: Tachycardia; Ventricular Tachycardia; Cardiac Arrhythmias; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Tachycardia; Tachycardia, Ventricular; Arrhythmias, Cardiac; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ICD/CRT-D with NIPS or EP Study — ICD/CRT-D implanted patients are tested for inducible MMVT during electrophysiology (EP) Study or Non-Invasive Programmed Stimulation (NIPS) Study

SUMMARY:
The intent of this observational study is to understand the role of non-invasive programmed stimulation (NIPS) to induce substrate based MMVT (Monomorphic Ventricular Tachycardia) in patients receiving new St. Jude Medical Implantable Cardioverter Defibrillator (ICD) or Cardiac Resynchronization Therapy Defibrillation (CRT-D) systems.

DETAILED DESCRIPTION:
Approximately 50 centers worldwide will participate in the study. Additional centers outside the US may be considered, as necessary. The anticipated enrollment duration is 48-60 months.

This study provides a mechanism for sites to refer subjects for potential enrollment to the Substrate Targeted Ablation Using the FlexAbility™ Ablation Catheter System for the Reduction of Ventricular Tachycardia (STAR-VT) Investigational Device Exemption (IDE) study (ClinicalTrials.gov NCT02130765).

Patients receiving ICD or CRT-D device implant (or have received it within 30 days) may be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

Patient is receiving a new SJM ICD or CRT-D implant system, which has study required programing capabilities and is appropriate for remote monitoring. Patients who have received the ICD or CRT-D up to 30 days prior to enrollment are also eligible.

Patient consents to have a NIPS/EP study.

Patient has documented Ejection Fraction (EF) < 50% and / or Right Ventricular (RV) dysfunction.

Patient has documented structural cardiomyopathy of any kind >1 month.

Patient is between 18 to 75 years of age.

Patient has been informed of the nature of the study and has agreed to its provisions and provided written informed consent using a form approved by the Institutional Review Board/Ethics Committee (IRB/EC).

Exclusion Criteria:

Patient has history of stroke.

Patient has had ST Segment elevation myocardial infarction (MI); or previous cardiac surgery within 60 days prior to enrollment.

Patient is pregnant or nursing.

Patient has chronic New York Heart Association (NYHA) Class IV heart failure.

Patient has limited life expectancy according to the investigator (less than one year).

Patient has had a recent coronary artery bypass graft (CABG) (< 60 days) or percutaneous coronary intervention (PCI) (< 30 days).

Patient is currently participating in an investigational drug or device study Patient is unable or unwilling to cooperate with the study procedures.

Patient has a prosthetic mitral or aortic valve.

Patient has mitral or aortic valvular heart disease requiring immediate surgical intervention.

Patient has Left Ventricular EF < 15%.

Patient has had a previous ablation procedure for ventricular tachycardia (VT), excluding remote (> 3 months) outflow tract tachycardia.

Patient has previously documented history of severe loss of kidney function or kidney failure.

Patient has premature ventricular contractions (PVC) or VT induced cardiomyopathy expected to resolve with ablation and will not require an ICD.

Patient has reversible cause of VT.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary study population includes patients who meet all inclusion/exclusion criteria, has had or will have market-approved St. Jude Medical ICD or CRT-D device systems implanted, and has no history of MMVT.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Rate of ICD/CRT-D implanted patients with documented monomorphic ventricular tachycardia. | 12 months

SECONDARY OUTCOMES:
Number of ICD shocks. | 12 months
Quality of Life via Short Form Survey (SF-36) | 12 months